CLINICAL TRIAL: NCT05155878
Title: Prognostic Factors, Operative Care and Short and Long Term Outcomes for Cysts and Tumors in Pancreas and the Periampullary Region
Brief Title: Prognostic Factors in Periampullary Tumors and Cysts
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Oskar Franklin, Principal Investigator, Umeå University
Other Study IDs: UmU-parpanc
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm; Pancreas Cyst; Pancreatic Fistula; Pancreas Disease; Bile Duct Cancer; Periampullary Cancer; Surgery; Surgery--Complications
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst; Pancreatic Fistula; Pancreatic Diseases; Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project aims at analysing prognostic and predictive factors involved in diagnostics and surgical treatment of cysts and tumors in the pancreas and periampullary region using both clinical data and blood and tissue samples for biomarker development and validation.

DETAILED DESCRIPTION:
From november 2021 an onward, study participants will be prospectively enrolled within the observational study. Before that, study participants are retrospectively enrolled. The study has a broad perspective including studies on clinical outcomes and prognostics based on patient and tumor characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Recommended surgery for tumor or cyst in the pancreas or periampullary region
* Information avalible in electronic journal files
* Informed consent (or deceased for retrospective part of the study)

Exclusion Criteria:

* No informed consent (and still alive at study initiation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have been recommended or already undergone surgery for a cyst or tumor in the pancreas or periampullary region
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Overall survival

SECONDARY OUTCOMES:
Complications | 10 years
  Clavien-Dindo, Specific procedure related outcomes
Radical resection | 10 years
  Rates of R0 vs R1/2 resections

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Franklin, MD/PhD, Principal Investigator — Umeå University Hospital
Locations (1):
- Surgical Clinic at Umeå University Hospital, Umeå, Sweden